CLINICAL TRIAL: NCT01337167
Title: A Phase III Randomized, Open-Label, Active-Comparator Controlled Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V419 in Infants When Given at 2, 4, and 6 Months Concomitantly With Prevnar 13™ and RotaTeq™
Brief Title: Safety, Tolerability, and Immunogenicity of V419 Given Concomitantly With Prevnar 13™ and RotaTeq™ (V419-005)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V419-005
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Bacterial Infections; Virus Diseases
Keywords: Diphtheria; Tetanus; Whooping Cough (pertussis); Poliomyelitis; Hepatitis B infection; Haemophilus influenzae type b infection
MeSH Terms: conditions — Bacterial Infections; Virus Diseases; Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Hepatitis B; Haemophilus Infections | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Haemophilus influenzae-type b polysaccharide-Neisseria meningitidis outer membrane protein conjugate vaccine; 13-valent pneumococcal vaccine; RotaTeq; Rotavirus Vaccines; pentacel; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- V419 (Experimental): V419 0.5 mL intramuscular injection (IM) at 2, 4, and 6 months of age; Daptacel™ 0.5 mL IM at 15 months of age; PedvaxHIB™ 0.5 mL IM at 15 months of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; and RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age.
  Interventions: Biological: V419; Biological: DAPTACEL™; Biological: PedvaxHIB™; Biological: Prevnar 13™; Biological: RotaTeq™
- Control (Active Comparator): Pentacel™ 0.5 mL IM at 2, 4, and 6 months of age; Recombivax HB vaccine 0.5 mL IM at 2 and 6 months of age; Daptacel™ 0.5 mL IM at 15 months of age; ActHIB™ 0.5 mL IM at 15 months of age; Prevnar 13™ 0.5 mL IM at 2, 4, 6, and 15 months of age; and RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age.
  Interventions: Biological: DAPTACEL™; Biological: Prevnar 13™; Biological: RotaTeq™; Biological: PENTACEL™; Biological: Recombivax HB vaccine; Biological: ActHIB™

INTERVENTIONS:
Biological: V419 — V419 (Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus, Haemophilus b Conjugate [Meningococcal Outer Membrane Protein Complex], and Hepatitis B [Recombinant] Vaccine) 0.5 mL intramuscular injection at 2, 4, and 6 months of age
  Arms: V419
Biological: DAPTACEL™ — DAPTACEL™ 0.5 mL intramuscular injection at 15 months of age
Biological: PedvaxHIB™ — PedvaxHIB™ 0.5 mL intramuscular injection at 15 months of age
  Arms: V419
Biological: Prevnar 13™ — Prevnar 13™ 0.5 mL intramuscular injection at 2, 4, 6, and 15 months of age
Biological: RotaTeq™ — RotaTeq™ 2 mL oral dose at 2, 4, and 6 months of age
  Other Names: V260
Biological: PENTACEL™ — PENTACEL™ 0.5 mL intramuscular injection at 2, 4, and 6 months of age
  Arms: Control
Biological: Recombivax HB vaccine — Recombivax HB vaccine 0.5 mL intramuscular injection at 2 and 6 months of age
  Arms: Control
Biological: ActHIB™ — ActHIB™ 0.5 mL intramuscular injection at 15 months of age
  Arms: Control

SUMMARY:
This is a study to assess the safety, tolerability, and immunogenicity of V419 (PR5I) when administered as an infant series at 2, 4, and 6 months of age followed by a toddler dose of DAPTACEL™, Prevnar 13™ and PedvaxHIB™ at 15 months of age. The study will determine whether subjects who receive V419 have a similar immune response to the vaccine compared to subjects who receive licensed component vaccine controls.

ELIGIBILITY:
Inclusion Criteria :

* Participant is a healthy infant
* Participant has received one dose of monovalent hepatitis B vaccine prior to or at 1 month of age

Exclusion Criteria :

* Participant has received more than one dose of monovalent hepatitis B vaccine or hepatitis B based combination vaccine prior to study entry
* Participant has been vaccinated with any acellular pertussis or whole cell pertussis based combination vaccines, haemophilus influenzae type b conjugate, poliovirus, pneumococcal conjugate or pneumococcal polysaccharide, rotavirus, or any combination of the above
* Participant has had a fever ≥38.0°C (≥110.4°F) within 24 hours of study enrollment
* Participant was vaccinated with any non-study vaccine (i.e., inactivated, conjugated, live virus vaccine) within 30 days prior to study enrollment, except for inactivated influenza vaccine which will be permitted 15 days or more prior to enrollment
* Participant has hepatitis B surface antigen (HBsAg) seropositivity (by medical history)
* Participant has a history of haemophilus influenzae type B, hepatitis B, diphtheria, tetanus, pertussis, poliomyelitis, rotavirus, or pneumococcal infection

Ages: 46 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1473 (Actual)
Dates: Start 2011-04-19 (Actual); Primary Completion 2013-05-09 (Actual); Study Completion 2013-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Marshall GS, Adams GL, Leonardi ML, Petrecz M, Flores SA, Ngai AL, Xu J, Liu G, Stek JE, Foglia G, Lee AW. Immunogenicity, Safety, and Tolerability of a Hexavalent Vaccine in Infants. Pediatrics. 2015 Aug;136(2):e323-32. doi: 10.1542/peds.2014-4102. PMID 26216331

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The infant series of vaccinations were those administered at 2, 4, and 6 months of age; the toddler vaccinations were those administered at 15 months of age. The Interim Period is the time between the last vaccination of the infant series and the time of administration of the toddler vaccination.
Period: Infant Series
Arm/Group | V419 | Control
Started | 986 | 487
Completed | 924 | 460
Not Completed | 62 | 27
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 13 | 7
Not completed — Non-compliance with study drug | 2 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 22 | 9
Not completed — Withdrawal by Subject | 15 | 4
Not completed — Randomized but not vaccinated | 5 | 3
Period: Interim Period
Arm/Group | V419 | Control
Started | 924 | 460
Completed | 843 | 420
Not Completed | 81 | 40
Not completed — Lost to Follow-up | 51 | 23
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Physician Decision | 6 | 3
Not completed — Protocol Violation | 5 | 3
Not completed — Withdrawal by Subject | 18 | 10
Not completed — Other protocol criterion not met | 0 | 1
Period: Toddler Vaccinations
Arm/Group | V419 | Control
Started | 843 | 420
Completed | 829 | 407
Not Completed | 14 | 13
Not completed — Lost to Follow-up | 11 | 12
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V419 | Control | Total
Number analyzed (Participants) | 986 | 487 | 1473
Age, Continuous [Mean (Standard Deviation); unit: Days] | 65.6 (7.5) | 65.0 (6.9) | 65.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 479 | 214 | 693
  Male | 507 | 273 | 780

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Responding to Polyribosylribitol Phosphate Antigen
Description: Participant serum samples were collected for testing with a radioimmunoassay for antibodies to Haemophilus influenza type b capsular polysaccharide polyribosylribitol phosphate. Response was evaluated for titer >=0.15 μg/mL and >=1.0 μg/mL.
Time Frame: Postdose 3 (Month 7)
Population: The analysis population included participants who met the inclusion criteria, were not protocol violators, had a vaccination window of 42 to 84 days after the previous dose, and a blood draw sample window for the endpoint of 28 to 51 days after dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 765 | 382
Percentage of participants
  Titer >=1.0 μg/mL | 84.97 [82.24 to 87.43] | 75.39 [70.76 to 79.63]
  Titer >=0.15 μg/mL | 97.25 [95.83 to 98.29] | 92.41 [89.28 to 94.86]
Statistical Analysis 1: Comparison: V419 vs Control; Non-inferiority for titer >=1.0 μg/mL; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 9.68, 95% CI 2-sided [4.83 to 14.83]
Statistical Analysis 2: Comparison: V419 vs Control; Non-inferiority for titer >=0.15 μg/mL; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 4.87, 95% CI 2-sided [2.23 to 8.14]
Statistical Analysis 3: Comparison: V419 vs Control; Secondary Analysis: Non-inferiority for titer >=0.15 μg/mL; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419-Ctrl) = 4.87, 95% CI 2-sided [2.23 to 8.14]

2. Primary Outcome: Percentage of Participants Responding to Hepatitis B Surface Antigen
Description: Participant serum samples were collected for testing with an enhanced chemiluminescence assay for antibodies to Hepatitis B Surface Antigen. Response was defined as a titer >=10 milli International units (mIU)/mL.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 688 | 353
Percentage of participants | 99.42 [98.52 to 99.84] | 98.58 [96.73 to 99.54]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 0.84, 95% CI 2-sided [-0.35 to 2.74]

3. Primary Outcome: Percentage of Participants Responding to Diphtheria Toxin
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to diphtheria toxin. Response was defined as a titer >=0.1 International unit (IU)/mL.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 786 | 393
Percentage of participants | 82.44 [79.60 to 85.04] | 86.26 [82.45 to 89.51]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p = 0.002, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = -3.84, 95% CI 2-sided [-8.02 to 0.66]

4. Primary Outcome: Percentage of Participants Responding to Tetanus Toxin
Description: Participant serum samples were collected for testing with an ELISA for anti-tetanus antibodies. Response was defined as a titer >=0.1 IU/mL.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 787 | 390
Percentage of participants | 99.87 [99.29 to 100.00] | 99.49 [98.16 to 99.94]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 0.39, 95% CI 2-sided [-0.28 to 1.74]

5. Primary Outcome: Percentage of Participants Responding to Pertussis Toxin
Description: Participant serum samples were collected for testing with an Enzyme-linked Immunosorbent Assay (ELISA) for antibodies to pertussis toxin. Response was defined as follows: 1) if the predose titer was <4 times the lower limit of quantitation (4X LLOQ) then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 796 | 391
Percentage of participants | 98.12 [96.91 to 98.94] | 98.47 [96.69 to 99.43]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = -0.33, 95% CI 2-sided [-1.80 to 1.60]

6. Primary Outcome: Percentage of Participants Responding to Pertussis Filamentous Hemagglutinin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis filamentous hemagglutinin. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 796 | 391
Percentage of participants | 87.31 [84.80 to 89.55] | 92.07 [88.93 to 94.55]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p = 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = -4.70, 95% CI 2-sided [-8.14 to -0.97]

7. Primary Outcome: Percentage of Participants Responding to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 794 | 390
Percentage of participants | 79.35 [76.36 to 82.11] | 82.05 [77.88 to 85.73]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = -2.67, 95% CI 2-sided [-7.27 to 2.23]

8. Primary Outcome: Percentage of Participants Responding to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae. Response was defined as follows: 1) if the predose titer was <4X LLOQ then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 796 | 391
Percentage of participants | 90.20 [87.92 to 92.18] | 86.19 [82.37 to 89.45]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 4.05, 95% CI 2-sided [0.23 to 8.28]

9. Primary Outcome: Percentage of Participants Responding to Poliovirus Type 1
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to Poliovirus Type 1. Response is defined as a titer >=8.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 806 | 398
Percentage of participants | 100.00 [99.54 to 100.00] | 98.24 [96.41 to 99.29]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 1.76, 95% CI 2-sided [0.85 to 3.59]
Statistical Analysis 2: Comparison: V419; Test type: Superiority or Other; p < 0.001, Clopper and Pearson; Acceptability requires that the lower bound of the 2-sided 95% CI of the response rate is >=90; Response Rate = 100.00, 95% CI 2-sided [99.54 to 100.00]

10. Primary Outcome: Percentage of Participants Responding to Poliovirus Type 2
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to Poliovirus Type 2. Response is defined as a titer >=8.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 801 | 399
Percentage of participants | 100.00 [99.54 to 100.00] | 99.75 [98.61 to 99.99]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 0.26, 95% CI 2-sided [-0.22 to 1.42]
Statistical Analysis 2: Comparison: V419; Test type: Superiority or Other; p < 0.001, Clopper and Pearson; Acceptability requires that the lower bound of the 2-sided 95% CI of the response rate is >=90; Response Rate = 100.00, 95% CI 2-sided [99.54 to 100.00]

11. Primary Outcome: Percentage of Participants Responding to Poliovirus Type 3
Description: Participant serum samples were collected for testing with a Micrometabolic Inhibition Test for neutralizing antibodies to Poliovirus Type 3. Response is defined as a titer >=8.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 790 | 396
Percentage of participants | 100.00 [99.53 to 100.00] | 99.75 [98.60 to 99.99]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -5%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 0.25, 95% CI 2-sided [-0.24 to 1.41]
Statistical Analysis 2: Comparison: V419; Test type: Superiority or Other; p < 0.001, Clopper and Pearson; Acceptability requires that the lower bound of the 2-sided 95% CI of the response rate is >=90; Response Rate = 100.00, 95% CI 2-sided [99.53 to 100.00]

12. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Toxin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis toxin. The unit of measure is ELISA units/mL (EU/mL).
Time Frame: Postdose 3 (Month 7)
Population: The analysis population included participants who met the inclusion criteria, were not protocol violators, had an infant vaccination window of 42 to 84 days after the previous dose, and a blood draw sample window for the endpoint of 28 to 51 days after dose 3.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 810 | 400
EU/mL | 110.40 [105.78 to 115.21] | 86.54 [81.87 to 91.48]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the Geometric Mean Concentration (GMC) ratio is >=0.67; p < 0.001, ANCOVA; GMC, GMC ratio, and p-value were adjusted for post- and prevaccination titer, vaccination group, and brand of birth dose of Hepatitis B vaccine; GMC Ratio (V419/Control) = 1.28, 95% CI 2-sided [1.20 to 1.38]

13. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Filamentous Hemagglutinin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis filamentous hemagglutinin.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 810 | 400
EU/mL | 48.17 [45.68 to 50.80] | 74.44 [68.99 to 80.33]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p = 0.786, ANCOVA; [statistical method as in outcome 12, analysis 1]; GMC Ratio (V419/Control) = 0.64, 95% CI 2-sided [0.59 to 0.70]

14. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 808 | 400
EU/mL | 56.22 [51.93 to 60.85] | 66.16 [59.50 to 73.57]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 12, analysis 1]; GMC Ratio (V419/Control) = 0.83, 95% CI 2-sided [0.73 to 0.95]

15. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 809 | 400
EU/mL | 235.62 [221.43 to 250.73] | 185.54 [169.33 to 203.31]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 12, analysis 1]; GMC Ratio (V419/Control) = 1.28, 95% CI 2-sided [1.15 to 1.42]

16. Primary Outcome: Percentage of Participants Responding to Pertussis Toxin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis toxin. Response was defined as follows: 1) if the predose titer was <4 times the lower limit of quantitation (4X LLOQ) then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 4 (Month 16)
Population: The analysis population included participants who met the inclusion criteria, were not protocol violators, had a vaccination window of 42 to 84 days after the previous dose, and a blood draw sample window for the endpoint of 28 to 51 days after dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 701 | 349
Percentage of participants | 99.29 [98.34 to 99.77] | 97.42 [95.16 to 98.81]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 1.88, 95% CI 2-sided [0.39 to 4.18]

17. Primary Outcome: Percentage of Participants Responding to Pertussis Filamentous Hemagglutinin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis filamentous hemagglutinin. Response was defined as follows: 1) if the predose titer was <4 times the lower limit of quantitation (4X LLOQ) then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 699 | 350
Percentage of participants | 94.42 [92.45 to 96.00] | 93.14 [89.97 to 95.56]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 1.30, 95% CI 2-sided [-1.67 to 4.78]

18. Primary Outcome: Percentage of Participants Responding to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin. Response was defined as follows: 1) if the predose titer was <4 times the lower limit of quantitation (4X LLOQ) then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 701 | 351
Percentage of participants | 93.01 [90.86 to 94.78] | 93.45 [90.33 to 95.80]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = -0.41, 95% CI 2-sided [-3.46 to 3.10]

19. Primary Outcome: Percentage of Participants Responding to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae. Response was defined as follows: 1) if the predose titer was <4 times the lower limit of quantitation (4X LLOQ) then the postdose titer was >=4X LLOQ; 2) if the predose titer was >=4X LLOQ then the postdose titer was >= the predose titer.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 700 | 351
Percentage of participants | 97.29 [95.79 to 98.36] | 91.17 [87.70 to 93.92]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 95% CI of the response rate difference is >= -10%; p < 0.001, Miettinen and Nurminen; Response rate, response rate difference and p-value were stratified by brand of birth dose of Hepatitis B vaccine; Response Rate Difference (V419 - Ctrl) = 6.18, 95% CI 2-sided [3.26 to 9.78]

20. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Toxin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis toxin.
Time Frame: Postdose 4 (Month 16)
Population: The analysis population included participants who met the inclusion criteria, were not protocol violators, had an infant vaccination window of 42 to 84 days after the previous dose, and a blood draw sample window for the endpoint of 28 to 51 days after dose 4.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 713 | 356
EU/mL | 127.22 [121.17 to 133.57] | 91.31 [85.09 to 97.98]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 12, analysis 1]; GMC Ratio (V419/Control) = 1.40, 95% CI 2-sided [1.28 to 1.52]

21. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Filamentous Hemagglutinin
Description: as for outcome 13
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 710 | 357
EU/mL | 88.92 [84.06 to 94.05] | 89.18 [82.54 to 96.35]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 12, analysis 1]; GMC Ratio (V419/Control) = 1.00, 95% CI 2-sided [0.91 to 1.10]

22. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Pertactin
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis pertactin.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 713 | 358
EU/mL | 108.05 [99.88 to 116.90] | 139.35 [124.81 to 155.58]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p = 0.014, ANCOVA; [statistical method as in outcome 12, analysis 1]; GMC Ratio (V419/Control) = 0.78, 95% CI 2-sided [0.68 to 0.89]

23. Primary Outcome: Geometric Mean Concentration of Antibodies to Pertussis Fimbriae
Description: Participant serum samples were collected for testing with an ELISA for antibodies to pertussis fimbriae.
Time Frame: Postdose 4 (Month 16)
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 713 | 358
EU/mL | 658.50 [617.53 to 702.20] | 414.66 [371.41 to 462.94]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 12, analysis 1]; GMC Ratio (V419/Control) = 1.58, 95% CI 2-sided [1.41 to 1.78]

24. Secondary Outcome: Geometric Mean Concentration of Antibodies to Polyribosylribitol Phosphate Antigen
Description: Participant serum samples were collected for testing with a radioimmunoassay for antibodies to Haemophilus influenza type b capsular polysaccharide polyribosylribitol phosphate.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 765 | 382
μg/mL | 5.11 [4.55 to 5.73] | 3.18 [2.66 to 3.81]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 12, analysis 1]; GMC Ratio (V419/Control) = 1.62, 95% CI 2-sided [1.32 to 1.98]

25. Secondary Outcome: Geometric Mean Concentration of Immunoglobulin A (IgA) Antibodies to Rotavirus
Description: Participant serum samples were collected for testing with an Enzyme-linked Immunosorbent assay for IgA antibodies to rotavirus.
Time Frame: Postdose 3 (Month 7)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: units/mL
Arm/Group | V419 | Control
Number analyzed (Participants) | 522 | 274
units/mL | 278.19 [246.99 to 313.32] | 274.46 [232.83 to 323.52]
Statistical Analysis 1: Comparison: V419 vs Control; Test type: Non-Inferiority or Equivalence — Non-inferiority requires that the lower limit of the 2-sided 95% CI of the GMC ratio is >=0.67; p < 0.001, ANCOVA; [statistical method as in outcome 12, analysis 1]; GMC Ratio (V419/Control) = 1.02, 95% CI 2-sided [0.83 to 1.24]

26. Secondary Outcome: Percentage of Participants Reporting Solicited Injection-site or Systemic Reactions
Description: Solicited injection-site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Pyrexia, Vomiting, Crying abnormal, Somnolence, Decreased appetite, and Irritability. Grade 3 Solicited injection site reaction: Pain, Cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling, >5 cm. Grade 3 Solicited systemic reactions: Pyrexia, >=39.5°C (>=103.1°F) rectal; Vomiting, >=6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal, >3 hours; Somnolence, Sleeping most of the time or difficult to wake up; Decreased appetite, Refuses >=3 feeds or refuses most feeds; Irritability, Inconsolable.
Time Frame: Up to 5 days after any infant vaccination (up to 6 months)
Population: Participants included in these analyses were All Subjects as Treated population and were defined as all vaccinated participants with safety follow up.
Measure: Number; unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 981 | 484
Percentage of participants
  Any injection-site pain | 73.4 | 71.8
  Grade 3 injection-site pain | 5.9 | 4.6
  Any injection-site erythema | 48.8 | 42.2
  Grade 3 injection-site erythema | 0.2 | 0.6
  Any injection-site swelling | 40.1 | 34.8
  Grade 3 injection-site swelling | 0.3 | 0.4
  Any pyrexia | 47.4 | 34.4
  Grade 3 pyrexia | 1.5 | 1.2
  Any vomiting | 25.7 | 21.5
  Grade 3 vomiting | 0.4 | 0.6
  Any crying abnormal | 74.8 | 72.3
  Grade 3 crying abnormal | 7.9 | 8.3
  Any somnolence | 74.1 | 71.6
  Grade 3 somnolence | 3.5 | 2.9
  Any decreased appetite | 48.9 | 43.3
  Grade 3 decreased appetite | 1.3 | 0.4
  Any irritability | 83.1 | 81.8
  Grade 3 irritability | 7.7 | 5.8

27. Secondary Outcome: Percentage of Participants Reporting One or More Solicited Adverse Events Related to Study Drug
Description: Solicited systemic adverse events: pyrexia, vomiting, crying abnormal, somnolence, decreased appetite, and irritability. Adverse events deemed related to study drug were those judged to be definitely related, probably related, or possibly related by the investigator.
Time Frame: Up to 5 days after any infant vaccination (up to 6 months)
Population: Participants included in this analyses were All Subjects as Treated population and were defined as all vaccinated participants with safety follow up.
Measure: Number; unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 981 | 484
Percentage of participants
  Any pyrexia | 45.1 | 32.1
  Any vomiting | 20.8 | 16.4
  Any crying abnormal | 71.4 | 68.5
  Any somnolence | 68.5 | 66.7
  Any decreased appetite | 45.7 | 40.2
  Any irritability | 79.6 | 77.4

28. Secondary Outcome: Percentage of Participants Reporting One or More Solicited Adverse Events Related to Study Drug
Description: as for outcome 27
Time Frame: Up to 5 days after each infant vaccination (up to 6 months)
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 981 | 484
Percentage of participants
  Any pyrexia, vaccination 1 | 16.1 | 12.6
  Any pyrexia, vaccination 2 (N=950, 472) | 26.6 | 16.4
  Any pyrexia, vaccination 3 (N=924, 460) | 26.6 | 16.2
  Any vomiting, vaccination 1 | 11.2 | 7.9
  Any vomiting, vaccination 2 (N=950, 472) | 10.2 | 8.5
  Any vomiting, vaccination 3 (N=924, 460) | 8.0 | 4.6
  Any crying abnormal, vaccination 1 | 50.9 | 48.7
  Any crying abnormal, vaccination 2 (N=950, 472) | 48.4 | 42.9
  Any crying abnormal, vaccination 3 (N=924, 460) | 42.0 | 36.1
  Any somnolence, vaccination 1 | 54.6 | 54.0
  Any somnolence, vaccination 2 (N=950, 472) | 42.9 | 41.4
  Any somnolence, vaccination 3 (N=924, 460) | 38.3 | 35.0
  Any decreased appetite, vaccination 1 | 27.4 | 24.0
  Any decreased appetite, vaccination 2 (N=950, 472) | 24.1 | 19.8
  Any decreased appetite, vaccination 3 (N=924, 460) | 20.9 | 17.3
  Any irritability, vaccination 1 | 63.2 | 60.5
  Any irritability, vaccination 2 (N=950, 472) | 56.6 | 52.7
  Any irritability, vaccination 3 (N=924, 460) | 52.7 | 48.8

29. Secondary Outcome: Percentage of Participants With Elevated Temperature by Severity
Description: Maximum temperature (all routes) was based on actual temperatures recorded with no adjustments to the measurement route. Maximum temperature (rectal) was required of all participants if the reading by another method was >=38.0°C.
Time Frame: Up to 5 days after any infant vaccination (up to 6 months)
Population: Participants included in this analyses were All Subjects as Treated population and were defined as all vaccinated participants with safety follow up and temperature data.
Measure: Number; unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 981 | 484
Percentage of participants
  All routes <38.0°C | 51.1 | 64.3
  All routes >=38.0°C and <38.5°C, mild | 24.2 | 19.1
  All routes >=38.5°C and <39.5°C, moderate | 22.7 | 15.5
  All routes >=39.5°C, severe | 2.0 | 1.1
  Rectal <38.0°C | 44.5 | 57.7
  Rectal >=38.0°C and <38.5°C, mild | 24.3 | 17.9
  Rectal >=38.5°C and <39.5°C, moderate | 21.6 | 14.9
  Rectal >=39.5°C, severe | 2.0 | 0.9
Statistical Analysis 1: Comparison: V419 vs Control; Estimated difference, all routes <38°C; Test type: Superiority or Other; Mean Difference (Final Values) = -13.1, 95% CI 2-sided [-18.4 to -7.7] — Mean Difference is V419 - Control. The 95% confidence intervals were based on the unstratified Miettinen and Nurminen method
Statistical Analysis 2: Comparison: V419 vs Control; Estimated difference, all routes >=38°C and <38.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 5.1, 95% CI 2-sided [0.5 to 9.5] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 3: Comparison: V419 vs Control; Estimated difference, all routes >=38.5°C and <39.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [2.8 to 11.2] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 4: Comparison: V419 vs Control; Estimated difference, all routes >=39.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.6 to 2.2] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 5: Comparison: V419 vs Control; Estimated difference, rectal <38°C; Test type: Superiority or Other; Mean Difference (Final Values) = -13.2, 95% CI 2-sided [-18.6 to -7.7] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 6: Comparison: V419 vs Control; Estimated difference, rectal >=38°C and <38.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 6.5, 95% CI 2-sided [1.9 to 10.8] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 7: Comparison: V419 vs Control; Estimated difference, rectal >=38.5°C and <39.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 6.7, 95% CI 2-sided [2.4 to 10.7] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 8: Comparison: V419 vs Control; Estimated difference, rectal >=39.5°C; Test type: Superiority or Other; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.3 to 2.4] — [estimate comment as in outcome 29, analysis 1]

30. Secondary Outcome: Percentage of Participants With Pyrexia, Febrile Convulsion, or Convulsion
Description: The percentage of participants with one or more adverse events (AE), serious adverse events (SAE), and vaccine-related SAE (pyrexia, febrile convulsion, and convulsion) is reported.
Time Frame: Up to 15 days after any infant vaccination (up to 6 months)
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 981 | 484
Percentage of participants
  Pyrexia AEs | 49.3 | 35.6
  Febrile convulsion AEs | 0 | 0
  Convulsion AEs | 0 | 0
  Pyrexia SAEs | 0 | 0
  Febrile convulsion SAEs | 0 | 0
  Convulsion SAEs | 0 | 0

31. Secondary Outcome: Percentage of Participants With Pyrexia, Febrile Convulsion, or Convulsion
Description: as for outcome 30
Time Frame: Up to 181 days after any infant vaccination (up to 12 months)
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | V419 | Control
Number analyzed (Participants) | 981 | 484
Percentage of participants
  Pyrexia SAEs | 0 | 0.2
  Febrile convulsion SAEs | 0.2 | 0
  Convulsion SAEs | 0.1 | 0.4
  Pyrexia vaccine-related SAEs | 0 | 0
  Febrile convulsion vaccine-related SAEs | 0 | 0
  Convulsion vaccine-related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs: up to 6 months after vaccination 3 (the last infant vaccination) and up to 15 days after vaccination 4 (the toddler vaccination); Vaccine-related SAEs and deaths: up to Month 16 (duration of the study); Other AEs: up to 15 days after any vaccination
Description: The All Subjects as Treated population included all randomized participants who received at least one dose of study vaccine and had safety follow-up
Arm/Group | V419 | Control
Serious Adverse Events (participants affected / at risk) | 58/980 | 32/483
Other Adverse Events (participants affected / at risk) | 939/980 | 458/483
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V419 (N=980) | Control (N=483)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Device expulsion (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 6 (6) | 5 (5)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 4 (5) | 3 (3)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Human herpesvirus 6 infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Meningitis enteroviral (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 6 (6) | 4 (4)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Roseola (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 12 (12) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Movement disorder (Nervous system disorders) | 0 (0) | 1 (1)
Tonic convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Kawasaki's disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V419 (N=980) | Control (N=483)
Diarrhoea (Gastrointestinal disorders) | 61 (68) | 22 (25)
Vomiting (Gastrointestinal disorders) | 282 (432) | 125 (186)
Crying (General disorders) | 788 (1933) | 370 (857)
Irritability (General disorders) | 853 (2389) | 415 (1109)
Pyrexia (General disorders) | 560 (1014) | 216 (356)
Otitis media (Infections and infestations) | 69 (76) | 26 (28)
Upper respiratory tract infection (Infections and infestations) | 100 (108) | 40 (41)
Decreased appetite (Metabolism and nutrition disorders) | 577 (1087) | 271 (469)
Somnolence (Nervous system disorders) | 755 (1863) | 369 (887)
Injection-site bruising (General disorders) | 62 (103) | 36 (61)
Injection-site erythema (General disorders) | 597 (2665) | 277 (1365)
Injection-site pain (General disorders) | 826 (4276) | 391 (2234)
Injection-site swelling (General disorders) | 513 (1974) | 219 (989)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/ presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.